CLINICAL TRIAL: NCT06752616
Title: Advancing the Quality of Treatment and Care for Acute Agitation in Emergency Psychiatry
Brief Title: Acute Agitation in Emergency Psychiatry
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Lone Baandrup (Other)
Collaborators: University Hospital Bispebjerg and Frederiksberg (Other); Capital Region's Pharmacy (Region Hovedstadens Apotek), Marielundvej 25, 2730 Herlev, Denmark (Unknown)
Responsible Party: Sponsor-Investigator, Lone Baandrup, Head of Clinic, clinical associate research professor, University of Copenhagen
Organization: University of Copenhagen (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-510201-18-00
Record Dates: First submitted 2024-12-22; First posted 2024-12-30 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Agitation
Keywords: Emergency psychiatry
MeSH Terms: conditions — Psychomotor Agitation | interventions — Lorazepam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Sublingual dexmedetomidine (Experimental)
  Interventions: Drug: Sublingual Dexmedetomidine
- Buccal midazolam (Experimental)
  Interventions: Drug: Buccal midazolam
- Oral lorazepam (Active Comparator)
  Interventions: Drug: Oral lorazepam

INTERVENTIONS:
Drug: Sublingual Dexmedetomidine — Sublingual dexmedetomidine 180 mcg, possible second dose 90 mcg after 2 hrs
  Arms: Sublingual dexmedetomidine
Drug: Buccal midazolam — Buccal midazolam 10 mg, possible second dose 10 mg after 2 hrs
  Arms: Buccal midazolam
Drug: Oral lorazepam — Oral lorazepam 4 mg, possible second dose 4 mg after 2 hrs
  Arms: Oral lorazepam

SUMMARY:
The purpose of the study is to improve the pharmacological treatment of psychiatric patients with acute agitation.

DETAILED DESCRIPTION:
The initial treatment of acute agitation aims to reduce suffering, abort the immediate risk of harm to self or others, and prevent the use of coercive measures such a physical and mechanical restraint. With this research project, we aim to build the initial structure of a visionary platform design and to examine the efficacy, tolerability, and safety of two hitherto under-investigated compounds versus the current standard of care for acutely agitated patients when de-escalation techniques have failed. After obtaining the results of the initial phase, we plan to apply for future funding to maintain and expand the platform design with the addition of relevant experimental arms. The proposed platform design aims to anwer the question What is the best treatment for acutely agitated patients in inpatient psychiatric settings?

ELIGIBILITY:
Inclusion Criteria:

* 18-64 years
* Agitation with the need for tranquillization in inpatient psychiatric settings including psychiatric emergency rooms
* Total score of ≥14 on the PANSS Excited Component (PEC)
* A score ≥4 on at least 1 of the 5 items of the PEC
* Informed consent obtained prior to the occurrence of the emergency

Exclusion Criteria:

* Involuntary psychiatric admission according to the Danish Mental Health Act
* Female patients who are breastfeeding
* Female patients aged <50 years and unable to perform a negative urine screen for pregnancy and not using safe contraceptives
* Body weight <50 kg
* Extreme obesity defined as estimated BMI≥ 40 kg/m2
* Clinical situations where acute administration of an antipsychotic is preferred to treat acute agitation (in the opinion of the investigator)
* The patient deemed unwilling or unable to cooperate with study procedures (in the opinion of the investigator)
* Insufficient language skills that interfere with reading, writing, and providing written informed consent in Danish or other available languages (in the opinion of the investigator)
* Clinical suspicion of contraindications for one of the treatment arms
* Use of benzodiazepines, other sedatives, or antipsychotic drugs in addition to usual treatment (i.e., additional PN sedative prescriptions) in the 4 hours before study treatment
* Known allergy to any of the study medications

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 132 (Estimated)
Dates: Start 2024-12-30 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
The Excited Component of the Positive and Negative Syndrome Scale (PEC) | 60 minutes
  The Excited Component of the Positive and Negative Syndrome Scale (PEC) consists of 5 clinician-rated items associated with agitation from the Positive and Negative Syndrome Scale (PANSS). Scores range from 5 to 35. Higher is worse.

SECONDARY OUTCOMES:
PEC score earliest time with difference | 30, 60, 90, and 120 minutes
  The earliest time where a statistically significant difference in agitation is apparent as measured by change from baseline PEC score (change from pre- to post-dose PEC score at 30, 60, 90, and 120 minutes)
Tranquillized or asleep | 30, 60, 90, and 120 minutes post-dose
  Proportion tranquillized or asleep (measured as ≤4 on the BARS**) by 30, 60, 90, and 120 minutes post-dose
Physical restraint | 12 hours post-dose
  Proportion physically restrained from administration to 12 hours post-dose
Mechanical restraint | 12 hours post-dose
  Proportion mechanically restrained from administration to 12 hours post-dose
Rescue medication | 4-12 hours post-dose
  Proportion given rescue medication 4-12 hours post-dose
Patient-reported satisfaction | From 2 to 24 hrs post-dose when the participant is able to cooperate
  Patient-reported satisfaction measured using 4 items from the Treatment Satisfaction Questionnaire for Medication II. Each item is answered on a 7-point Likert scale from 1 (extremely dissatisfied) to 7 (extremely satisfied). Score range is from 4 to 28. Higher is better.

CONTACTS AND LOCATIONS:
Overall Officials: Lone Baandrup, MD, DMSc, Principal Investigator — Mental Health Center Copenhagen
Locations (1):
- Mental Health Center Copenhagen, Bispebjerg, Copenhagen N, Denmark

IPD SHARING:
Plan to Share IPD: Yes
The study protocol will be available in the CTIS. After publication of primary and secondary outcomes, IPD will be handed over to the Danish National Archives where data will be archived for 25 years. IPD will be shared upon reasonable reuqest after publication of primary and secondary outcomes.